CLINICAL TRIAL: NCT02947321
Title: GREAT Knee Pain Reduction Trial, Genicular Radiofrequency Ablation Efficacy in Achieving Total Knee Pain Reduction Trial
Brief Title: Genicular Radiofrequency Ablation Efficacy in Achieving Total Knee Pain Reduction Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Puneet Mishra, Assistant Professor of Anesthesiology and Pain Medicine, BH Robbins Scholar, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160663
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Knee Arthroplasty, Total; Osteoarthritis; Radiologic Tibiofemoral Osteoarthritis
Keywords: Radiofrequency ablation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA Group (Experimental): A genicular nerve RFA will be performed prior to planned total knee arthroplasty.
  Interventions: Procedure: Genicular Nerve RFA
- Control Group (Sham Comparator): A sham genicular nerve RFA will be performed prior to planned total knee arthroplasty.
  Interventions: Procedure: Sham Genicular Nerve RFA

INTERVENTIONS:
Procedure: Genicular Nerve RFA — Under fluoroscopic guidance, the target locations based on boney landmarks of the superior lateral (SL), superior medial (SM), and inferior medial (IL) branches of the genicular nerve will be determined. RFA probes will be placed and connected to the RFA generator and the generator is activated. The RFA is performed.
  Arms: RFA Group
Procedure: Sham Genicular Nerve RFA — Under fluoroscopic guidance, the target locations based on boney landmarks of the superior lateral (SL), superior medial (SM), and inferior medial (IL) branches of the genicular nerve will be determined. The RFA probes for the control group will not be connected to the RFA generator (no neurotomy); however, the generator will still be activated to mimic the RFA group.
  Arms: Control Group

SUMMARY:
Given the benefits of genicular nerve radiofrequency ablation (RFA) in improving pain and functional status in non-surgical patients with knee osteoarthritis as well as the high prevalence of postoperative pain from total knee arthroplasty (TKA), this study is designed to determine the efficacy of preoperative genicular nerve RFA in improving acute and chronic postoperative pain as well as functional status in patients undergoing TKA. Patients will be randomized to one of two study arms: RFA group (genicular nerve thermal RFA) or control group (RFA needles placed in proper location without effective neurotomy).

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a common and effective treatment for severe knee osteoarthritis. As the average age of the population increases in developed countries, the number of TKAs performed is projected to increase to 3.48 million procedures per year by 2030, a 673% increase from 2005. Although TKA is widely accepted as an efficacious form of treatment for severe knee osteoarthritis, the incidence of patient dissatisfaction and postoperative pain cannot be ignored. Genicular nerve RFA has been performed in non-surgical patients with chronic knee osteoarthritis with significant post procedure improvement in pain and functional status. This study is designed to determine the efficacy of preoperative genicular nerve RFA in improving acute and chronic postoperative pain as well as functional status in patients undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for total knee arthroplasty secondary to osteoarthritis
* Radiologic tibiofemoral osteoarthritis (Kellgren-Lawrence grade 2-4)

Exclusion Criteria:

* Worst knee pain score on day of evaluation <4/10
* Already taking opioids >100 mg/day of morphine equivalent dose
* Infectious etiology (over RFA insertion site or systemic)
* Workers compensation
* History of adverse reaction to local anesthetic or contrast
* History of intraarticular injection in the last 6 weeks with steroids or hyaluronic acids
* Prior total knee arthroplasty
* Prior open knee surgery or ligament reconstruction
* Prior RFA of knee joint
* Connective tissue diseases affecting the knee
* Sciatic pain
* Pacemaker
* Pregnancy
* Severe medical disease
* Serious neurological disorders
* Serious psychiatric disorders
* Suicidal or homicidal ideation
* BMI>50

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Comparison of pain score at rest | On the day of genicular nerve RFA or sham procedure, preoperatively on the day of surgery, on postoperative day 1 and 2, and at week 2, 6, 24, and 52.
  Pain score at rest using an 11-point Pain Intensity Numerical Rating Scale (PI-NRS)
Comparison of pain score with ambulation | On the day of genicular nerve RFA or sham procedure, preoperatively on the day of surgery, on postoperative day 1 and 2, and at week 2, 6, 24, and 52.
  Pain score with ambulation using an 11-point Pain Intensity Numerical Rating Scale (PI-NRS)

SECONDARY OUTCOMES:
Comparison of PROMIS physical function score | On the day of genicular nerve RFA or sham procedure, preoperatively on the day of surgery, and at week 2, 6, 24, and 52
  Physical function assessment using the PROMIS physical function score
Comparison of PROMIS global health score | On the day of genicular nerve RFA or sham procedure, preoperatively on the day of surgery, and at week 2, 6, 24, and 52
  Global health assessment using the PROMIS global health score
Comparison of Knee Injury and Osteoarthritis Outcome Joint Replacement Score (KOOS JR) | On the day of genicular nerve RFA or sham procedure, preoperatively on the day of surgery, and at week 2, 6, 24, and 52
  Outcome assessment using the Knee Injury and Osteoarthritis Outcome Joint Replacement Score (KOOS JR)
Comparison of 7-point Patient Global Impression of Change (PGIC) | Preoperatively on the day of surgery, and at week 2, 6, 24, and 52
  Assessment of the subject's belief about the efficacy of treatment using the PGIC.
Comparison of Mobility using Timed Up and Go Test (TUG) | Day of genicular RFA or sham procedure, and postoperative day 1
  Assessment of mobility using the TUG test
Comparison of Depression assessment using Center for Epidemiologic Studies Depression Scale (CES-D) | Day of genicular RFA or sham procedure and at 6 weeks postoperatively
  Screening for depression using the CES-D
Comparison of Total opioid use in morphine equivalents | Day of genicular RFA or sham procedure, day of surgery, post op dy 1 and 2, and at weeks 2,6 postoperatively
Assessment of pain location using Michigan Body Map | Day of genicular nerve RFA
Assessment of pain catastrophizing using Catastrophizing General Chronic Pain (CAT) Scale | Day of genicular RFA or sham procedure
Comparison of quadriceps strength | Day of genicular RFA or sham procedure, and at weeks 2 and 6 postoperatively
Comparison Range of Motion - Knee | Day of genicular RFA or sham procedure, and at weeks 2 and 6 postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Mishra, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597-606. doi: 10.1056/NEJMoa1505467. PMID 26488691
- [Background] Singh JA, Vessely MB, Harmsen WS, Schleck CD, Melton LJ 3rd, Kurland RL, Berry DJ. A population-based study of trends in the use of total hip and total knee arthroplasty, 1969-2008. Mayo Clin Proc. 2010 Oct;85(10):898-904. doi: 10.4065/mcp.2010.0115. Epub 2010 Sep 7. PMID 20823375
- [Background] Lenguerrand E, Wylde V, Gooberman-Hill R, Sayers A, Brunton L, Beswick AD, Dieppe P, Blom AW. Trajectories of Pain and Function after Primary Hip and Knee Arthroplasty: The ADAPT Cohort Study. PLoS One. 2016 Feb 12;11(2):e0149306. doi: 10.1371/journal.pone.0149306. eCollection 2016. PMID 26871909
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Singh JA, Lewallen DG. Are outcomes after total knee arthroplasty worsening over time? A time-trends study of activity limitation and pain outcomes. BMC Musculoskelet Disord. 2014 Dec 17;15:440. doi: 10.1186/1471-2474-15-440. PMID 25519240
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Wylde V, Dieppe P, Hewlett S, Learmonth ID. Total knee replacement: is it really an effective procedure for all? Knee. 2007 Dec;14(6):417-23. doi: 10.1016/j.knee.2007.06.001. Epub 2007 Jun 26. PMID 17596949
- [Background] Grosu I, Lavand'homme P, Thienpont E. Pain after knee arthroplasty: an unresolved issue. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1744-58. doi: 10.1007/s00167-013-2750-2. Epub 2013 Nov 8. PMID 24201900
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Dunbar MJ, Richardson G, Robertsson O. I can't get no satisfaction after my total knee replacement: rhymes and reasons. Bone Joint J. 2013 Nov;95-B(11 Suppl A):148-52. doi: 10.1302/0301-620X.95B11.32767. PMID 24187375
- [Background] Wylde V, Hewlett S, Learmonth ID, Dieppe P. Persistent pain after joint replacement: prevalence, sensory qualities, and postoperative determinants. Pain. 2011 Mar;152(3):566-572. doi: 10.1016/j.pain.2010.11.023. Epub 2011 Jan 15. PMID 21239114
- [Background] Wylde V, Rooker J, Halliday L, Blom A. Acute postoperative pain at rest after hip and knee arthroplasty: severity, sensory qualities and impact on sleep. Orthop Traumatol Surg Res. 2011 Apr;97(2):139-44. doi: 10.1016/j.otsr.2010.12.003. Epub 2011 Mar 8. PMID 21388906
- [Background] Srikandarajah S, Gilron I. Systematic review of movement-evoked pain versus pain at rest in postsurgical clinical trials and meta-analyses: a fundamental distinction requiring standardized measurement. Pain. 2011 Aug;152(8):1734-1739. doi: 10.1016/j.pain.2011.02.008. Epub 2011 Mar 12. PMID 21402445
- [Background] Puolakka PA, Rorarius MG, Roviola M, Puolakka TJ, Nordhausen K, Lindgren L. Persistent pain following knee arthroplasty. Eur J Anaesthesiol. 2010 May;27(5):455-60. doi: 10.1097/EJA.0b013e328335b31c. PMID 20299989
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Karaman H, Tufek A, Kavak GO, Yildirim ZB, Uysal E, Celik F, Kaya S. Intra-articularly applied pulsed radiofrequency can reduce chronic knee pain in patients with osteoarthritis. J Chin Med Assoc. 2011 Aug;74(8):336-40. doi: 10.1016/j.jcma.2011.06.004. Epub 2011 Jul 23. PMID 21872812
- [Derived] Mishra P, Edwards D, Huntoon M, Sobey C, Polkowski G, Corey J, Mishra KL, Shinar A, Engstrom S, Palmer C, Bruehl S. Is preoperative genicular radiofrequency ablation effective for reducing pain following total knee arthroplasty? A pilot randomized clinical trial. Reg Anesth Pain Med. 2021 Sep;46(9):752-756. doi: 10.1136/rapm-2021-102501. Epub 2021 Jul 2. PMID 34215667